CLINICAL TRIAL: NCT07338123
Title: A Randomized Controlled Trial (RCT) of Yiqi Huoxue Jiedu Formula Combined With Bacteriophages in the Treatment of Severe Pneumonia Caused by Drug-resistant Gram-negative Bacilli
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Chief Physician, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025ZD0549303
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- YHDF Placebo + Bacteriophage Placebo Group (Placebo Comparator)
  Interventions: Drug: YHDF Placebo; Drug: Bacteriophage Placebo
- YHDF Placebo + Bacteriophage Group (Placebo Comparator)
  Interventions: Drug: YHDF Placebo; Drug: Bacteriophage
- YHDF Drug + Bacteriophage Placebo Group (Placebo Comparator)
  Interventions: Drug: YHDF Drug; Drug: Bacteriophage Placebo
- YHDF Drug + Bacteriophage Group (Experimental)
  Interventions: Drug: YHDF Drug; Drug: Bacteriophage

INTERVENTIONS:
Drug: YHDF Drug — 7-day treatment with YHDF Drug
  Arms: YHDF Drug + Bacteriophage Group; YHDF Drug + Bacteriophage Placebo Group
Drug: YHDF Placebo — 7-day treatment with YHDF placebo
  Arms: YHDF Placebo + Bacteriophage Group; YHDF Placebo + Bacteriophage Placebo Group
Drug: Bacteriophage — 7-14-day treatment with phage
  Arms: YHDF Drug + Bacteriophage Group; YHDF Placebo + Bacteriophage Group
Drug: Bacteriophage Placebo — 7-14-day treatment with phage placebo
  Arms: YHDF Drug + Bacteriophage Placebo Group; YHDF Placebo + Bacteriophage Placebo Group

SUMMARY:
Through a prospective randomized controlled trial, we systematically evaluate the effects of Yiqi Huoxue Jiedu Formula combined with bacteriophage therapy on the bacterial clearance rate, disease improvement rate and mortality rate in patients with severe pneumonia caused by drug-resistant bacteria, so as to clarify its clinical transformation value.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria for severe pneumonia caused by drug-resistant Gram-negative bacilli and conform to the TCM syndrome differentiation of Qi deficiency, toxin accumulation and blood stasis syndrome; patients confirmed by rapid on-site microbiological evaluation (M-ROSE), clinical microbial culture and drug susceptibility testing (based on the drug susceptibility test results of our hospital or other Grade A tertiary hospitals) to be infected with multidrug-resistant Klebsiella pneumoniae, Acinetobacter baumannii or Pseudomonas aeruginosa; aged 18 to 85 years old; patients or their family members agree to cooperate with the collection of upper and lower respiratory tract specimens, consent to bronchoscopy plus bronchoalveolar lavage, and agree to receive nebulized inhalation of bacteriophage therapy; patients or their family members have fully read, understood and signed the informed consent form.

Exclusion Criteria:

* Women who are pregnant or lactating; patients with immunodeficiency; patients receiving immunosuppressive therapy or suffering from immunodeficiency diseases; patients who have received mechanical ventilation for more than 60 days prior to enrollment; patients with active pulmonary tuberculosis, lung abscess, or Grade D chronic obstructive pulmonary disease (COPD); patients with incomplete sampling or clinical data; patients with known allergies to bacteriophage products or the components of Yiqi Huoxue Jiedu Formula; patients judged by the researchers as unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Clearance rate of drug-resistant bacteria | 14 days

SECONDARY OUTCOMES:
Time to clinical improvement | 7 days
All-cause mortality | 28 days

IPD SHARING:
Plan to Share IPD: Undecided